CLINICAL TRIAL: NCT02412020
Title: Treatment of Chronic Idiopathic Cough and Chronic Cough in Patients With Idiopathic Pulmonary Fibrosis With PA101
Brief Title: Treatment of Refractory Chronic Cough With PA101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patara Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA101-CC-02
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA101 (Experimental): PA101, 40 mg administered via inhalation three times daily for 14 days
  Interventions: Drug: PA101; Drug: Placebo
- Placebo (Placebo Comparator): Placebo PA101, administered via inhalation three times daily for 14 days
  Interventions: Drug: PA101; Drug: Placebo

INTERVENTIONS:
Drug: PA101
Drug: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, 2-period crossover, 2-cohort study in adult patients with refractory chronic cough.

The purpose of the study is to assess the efficacy and safety of inhaled PA101 delivered via eFlow high efficiency nebulizer for treating refractory chronic cough.

DETAILED DESCRIPTION:
The study consists of 2 treatment cohorts with refractory chronic cough: Idiopathic Pulmonary Fibrosis (IPF, Cohort 1) and Chronic Idiopathic Cough (CIC, Cohort 2). In each cohort, the study will include two treatment periods of 14 days each separated by a Washout Period of 14 days between Period 1 and Period 2. The two periods will be identical except that in Period 2, patients will crossover to the alternate treatment from that received in Period 1, according to a 1:1 randomization scheme.

During each period, patients will self-administer study drug (i.e., 40 mg PA101 or Placebo PA101 via eFlow) three times daily for 14 consecutive days of each period. Objective cough count will be recorded over 24-hour period using a cough count device (Leicester Cough Monitor) at the Baseline, Day 7 and Day 14 of each treatment period.

In the IPF cohort, patients will be allowed to use antifibrotic therapy (i.e., pirfenidone, nintedanib, and N-acetylcysteine) during the course of the study provided that the dose is stabilized at least 3 months prior to Screening and throughout the study period.

Clinical safety assessments will be performed at the start and end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Pulmonary Fibrosis (based on presence of definitive or possible usual interstitial pneumonia UIP pattern on high-resolution computed tomography and after excluding lung diseases associated with environmental and occupational exposure, with connective tissue disease and with drugs; transfer capacity for carbon monoxide corrected for hemoglobin [TLCOc] >25% predicted within 12 months of Screening; and forced vital capacity [FRC] >50% predicted within 1 month of Screening) or Chronic Idiopathic Cough (that is unresponsive to targeted treatment for identified underlying triggers including post-nasal drip, asthmatic/non-asthmatic eosinophilic bronchitis, and gastro-esophageal reflux disease)
* Refractory chronic cough for at least 8 weeks
* Daytime cough severity score >40 mm on Cough Severity VAS at Screening
* Daytime average cough count ≥15 per hour at Screening
* Willing and able to provide written informed consent

Exclusion Criteria:

* Current or recent history of clinically significant medical condition, laboratory abnormality or illness that could put the patient at risk or compromise the quality of the study data as determined by the investigator
* Upper or lower respiratory tract infection within 4 weeks of Screening
* History of malignancy treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma or cervix carcinoma in situ
* Current or recent history (within 12 months) of excessive use or abuse of alcohol
* Current or recent history (within 12 months) of abusing legal drugs or use of illegal drugs or substances
* Participation in any other investigational drug study within 4 weeks of Screening
* Use of prednisone, narcotic antitussives, baclofen, gabapentin, inhaled corticosteroids, benzonatate, dextromethorphan, carbetapentane, H1 antihistamines, leukotriene modifiers, and cromolyn sodium within 2 weeks of Screening
* Pregnant or breastfeeding females, or if of child-bearing potential unwilling to practice acceptable means of birth control or abstinence during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
cough frequency | 14 days
  objective 24-hour cough monitoring

SECONDARY OUTCOMES:
cough severity | 14 days
  VAS scale for cough severity
cough-related quality of life | 14 days
  Leicester Cough Questionnaire

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - Isala, Zwolle
- United Kingdom (5):
  - Hull Clinical Trials Unit, Cottingham, East Yorkshire
  - Uni Hospital Leicester, Leicester
  - King's College Hospital, London
  - Royal Brompton & Harefield Hospital, London
  - Uni Hospital North Staffordshire, Stoke-on-Trent

REFERENCES:
- [Derived] Birring SS, Wijsenbeek MS, Agrawal S, van den Berg JWK, Stone H, Maher TM, Tutuncu A, Morice AH. A novel formulation of inhaled sodium cromoglicate (PA101) in idiopathic pulmonary fibrosis and chronic cough: a randomised, double-blind, proof-of-concept, phase 2 trial. Lancet Respir Med. 2017 Oct;5(10):806-815. doi: 10.1016/S2213-2600(17)30310-7. Epub 2017 Sep 8. PMID 28923239